CLINICAL TRIAL: NCT06163248
Title: Effect of a Chrono Nutrition Intervention on Insulin Resistance in Adults With Type 2 Diabetes
Brief Title: Chrono Nutrition and Insulin Resistance in Diabetes
Acronym: Chrono
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4494
Record Dates: First submitted 2023-10-05; First posted 2023-12-08 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Chrono nutrition; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Chrono nutrition intervention:
  Participants will be asked to fast for 12 hours each day. During the fasting period, they may consume non-caloric beverages such as plain water, coffee or unsweetened tea. They will be asked to follow a dietary plan in which the total daily calorie intake will be calculated using indirect calorimetry, subtracting 500 calories from the total calorie amount. The dietary plan will have the following macronutrient distribution: 40% carbohydrates (<10% simple carbohydrates), 20% protein, and 40% fats (6-11% polyunsaturated, 15-20% monounsaturated, and <10% saturated). The plan will consist of 3 meals: breakfast will account for 40% of the total calories. Dinner will include only 10% of the total grams of carbohydrates. The order of food consumption should be: 1) vegetables, 2) proteins, 3) complex carbohydrates, and 4) simple carbohydrates (fruits).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chrono nutrition (Experimental): 1. During the 6-month period, participants will be asked to fast for 12 hours each day. During the fasting period, they may consume non-caloric beverages such as plain water, coffee, or unsweetened tea.
  2. The total daily calorie intake will be calculated using indirect calorimetry, considering the participant's current weight, age, sex, and physical activity level. 500 calories will be subtracted from the total calorie amount.
  3. The dietary plan will have the following macronutrient distribution: 40% carbohydrates (<10% simple carbohydrates), 20% protein, and 40% fats (6-11% polyunsaturated, 15-20% monounsaturated, and <10% saturated).
  4. The plan will consist of 3 meals and breakfast will account for 40% of the total calories.
  5. During dinner, only 10% of the total grams of carbohydrates will be included.
  6. The order of food consumption should be as follows: 1) vegetables, 2) proteins, 3) complex carbohydrates, and 4) simple carbohydrates (fruits).
  Interventions: Other: Chrono nutrition
- Standard (Active Comparator): 1. The total daily calorie intake will be calculated using indirect calorimetry, considering the participant's current weight, age, sex, and physical activity level. 500 calories will be subtracted from the total calorie amount.
  2. The dietary plan will have the following macronutrient distribution: 40% carbohydrates (<10% simple carbohydrates), 20% protein, and 40% fats (6-11% polyunsaturated, 15-20% monounsaturated, and <10% saturated).
  3. The plan will consist of 3 meals with an isocaloric distribution, with each meal containing 33% of the total calories.
  Interventions: Other: Standard

INTERVENTIONS:
Other: Chrono nutrition — An integral nutritional strategy involving timing, order and distribution of macronutrients
  Arms: Chrono nutrition
Other: Standard — Conventional nutritional strategy involving isocaloric distribution with no specific timing
  Arms: Standard

SUMMARY:
The goal of this randomized clinical trial is to determine the effect of a chrono nutrition intervention compared with a usual dietary intervention on insulin resistance in individuals with type 2 diabetes with overweight or obesity over a 6-month period.

The main question it aims to answer is: What is the effect of a chrono nutrition intervention compared to a standard intervention on insulin resistance in individuals with T2D (type 2 diabetes) with overweight or obesity over a 6-month period?

Participants:

* Will be asked to fast for 12 hours each day. During the fasting period, they may consume non-caloric beverages such as plain water, coffee, or unsweetened tea.
* They will be asked to follow a dietary plan in which the total daily calorie intake will be calculated using indirect calorimetry, subtracting 500 calories from the total calorie amount.
* The dietary plan will have the following macronutrient distribution: 40% carbohydrates (<10% simple carbohydrates), 20% protein, and 40% fats (6-11% polyunsaturated, 15-20% monounsaturated, and <10% saturated).
* The plan will consist of 3 meals: breakfast will account for 40% of the total calories. Dinner will include only 10% of the total grams of carbohydrates.
* The order of food consumption should be: 1) vegetables, 2) proteins, 3) complex carbohydrates, and 4) simple carbohydrates (fruits).

Researchers will compare the chrono nutrition strategy with a standard dietary intervention to see the effect in insulin resistance.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is considered one of the main public health problems. During the last decade the incidence of T2D has increased exponentially leading to an increased incidence in cardiovascular disease, premature death, blindness and non-traumatic limb amputation. Novel therapeutic interventions have become imperative.

Dietary interventions are the cornerstone in managing and preventing T2D, however there is heterogeneity in the interventions and approaches currently available. The main objective of a dietary intervention is modest weight reduction achieved through calorie deficit and reduction in the consumption of carbohydrates and fats. Dietary interventions with a chrono nutrition focus establish an eating regime with calorie and macronutrient distribution taking into account sleeping and fasting hours, which are associated with metabolic alterations. This approach looks beyond calorie deficit and weight loss as primary outcomes.

Nutrition, physical activity, and education are fundamental pillars for achieving metabolic control in T2D. It is well-described that a nutritional treatment alone can improve glycemic control and the quality of life of patients. It is interesting to note that the timing of meals throughout the 24-hour period seems to play an important role, similar to the number of meals per day or the total calorie intake. Furthermore, the daily pattern of fasting-feeding is influenced by the sleep-wake cycle pattern, which is one of the most evident adaptations to circadian rhythms and plays a significant role in maintaining optimal health.

Interventions targeting aspects such as food type, meal timing, quality, and quantity can be a simple and promising strategy that can positively or negatively impact metabolic health, regardless of body weight modification. This evidence supports chrono nutrition as a novel strategy in the field of nutrition, primarily focusing on studying the interaction between nutrition, feeding, and the circadian rhythm. The implementation of new nutritional strategies based on circadian rhythms contributes to improving adherence to dietary treatment and preventing potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes (T2D)
* HbA1c < 8.5%
* BMI ≥ 25 kg/m2 and < 35 kg/m2
* Stable pharmacological treatment for the last 3 months
* Willingness to participate in the protocol.

Exclusion Criteria:

* Insulin treatment
* Hospitalization in the previous three months
* Disease with adverse prognosis (SIDA, cancer)
* Rheumatologic diseases under immunosuppressive treatment (SLE, RA)
* Acute infection or febrile syndrome
* Hepatic cirrhosis
* Glomerular filtration rate <60 ml/min
* Other diabetes types (LADA, T1, MODY)
* Fasting triglycerides >500 mg/dl
* Pregnancy
* Lactation
* Steroid treatment
* High performance athletes
* Estrogen treatment
* Weight reduction >5% in the last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in insulin resistance (M value) | Six months
  Change in insulin resistance (M value) assessed with an euglycemic-hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Change in visceral adipose (liters) | Six months
  Change in visceral adipose tissue amount
Change in glycated hemoglobin (%) | Six months
  Change in glycated hemoglobin
Change in lipid profile (mg/dl) | Six months
  Change in lipid profile

OTHER OUTCOMES:
Change in hepatic steatosis and fibrosis (decibels and kilopascals) | Six months
  Change in hepatic steatosis and fibrosis assessed with elastography
Hunger and satiety (score) | Six months
  Change in hunger and satiety assessed with visual analog scale for hunger and satiety

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

REFERENCES:
- [Background] Henry CJ, Kaur B, Quek RYC. Chrononutrition in the management of diabetes. Nutr Diabetes. 2020 Feb 19;10(1):6. doi: 10.1038/s41387-020-0109-6. PMID 32075959
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Beneficial metabolic effects of regular meal frequency on dietary thermogenesis, insulin sensitivity, and fasting lipid profiles in healthy obese women. Am J Clin Nutr. 2005 Jan;81(1):16-24. doi: 10.1093/ajcn/81.1.16. PMID 15640455
- [Background] Stote KS, Baer DJ, Spears K, Paul DR, Harris GK, Rumpler WV, Strycula P, Najjar SS, Ferrucci L, Ingram DK, Longo DL, Mattson MP. A controlled trial of reduced meal frequency without caloric restriction in healthy, normal-weight, middle-aged adults. Am J Clin Nutr. 2007 Apr;85(4):981-8. doi: 10.1093/ajcn/85.4.981. PMID 17413096
- [Background] Lopez-Minguez J, Saxena R, Bandin C, Scheer FA, Garaulet M. Late dinner impairs glucose tolerance in MTNR1B risk allele carriers: A randomized, cross-over study. Clin Nutr. 2018 Aug;37(4):1133-1140. doi: 10.1016/j.clnu.2017.04.003. Epub 2017 Apr 10. PMID 28455106
- [Background] Jakubowicz D, Wainstein J, Landau Z, Ahren B, Barnea M, Bar-Dayan Y, Froy O. High-energy breakfast based on whey protein reduces body weight, postprandial glycemia and HbA1C in Type 2 diabetes. J Nutr Biochem. 2017 Nov;49:1-7. doi: 10.1016/j.jnutbio.2017.07.005. Epub 2017 Jul 21. PMID 28863364